CLINICAL TRIAL: NCT04314219
Title: Comparing Post-Transplant Cyclophosphamide with Calcineurin Inhibitors As a GVHD Prophylaxis to Standard Care of Methotrexate and Calcineurin Inhibitors for Acute Leukemia Incorporating Patient Pharmacogenomics Profiling
Brief Title: Comparing Post-Transplant Cyclophosphamide As GVHD Prophylaxis to Standard of Care for Acute Leukemia Patients
Acronym: PTCy-PMAT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2181104; Saudi FDA (Other: 19052902)
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-10

CONDITIONS: Acute Lymphoblastic Leukemia (ALL) in Complete Remission; Acute Myeloid Leukemia (AML) in Remission
Keywords: Sibling Donor Transplant; Allogeneic hematopoietic cell transplantation; GvHD Prophylaxis; Myeloablative regimen
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Pathologic Complete Response; Leukemia, Myeloid, Acute | interventions — Cyclophosphamide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Intervention (Experimental): Peripheral blood matched related donor HCT, using myeloablative conditioning regimen (IV Busulfan/IV Fludarabine for AML, IV VP16/TBI for ALL) HCT with cyclophosphamide, and oral tacrolimus (or another calcineurin inhibitor if intolerant for tacrolimus) for GVHD prophylaxis. Cyclophosphamide will be given at a dose of 50 mg/kg/day IV on Day +3 and Day +5 post stem cell infusion (only 2 doses).
  Interventions: Drug: Cyclophosphamide 50mg
- Arm 2: Standard of Care (Active Comparator): Peripheral blood matched related donor HCT, using myeloablative conditioning regimen (IV Busulfan/IV Fludarabine for AML, IV VP16/TBI for ALL) HCT with methotrexate, and oral tacrolimus (or another calcineurin inhibitor if intolerant for tacrolimus) for GVHD prophylaxis
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Cyclophosphamide 50mg — Cyclophosphamide as GVHD prophylaxis will be on day +3 and day +5
  Arms: Arm 1: Intervention
Drug: Methotrexate — Methotrexate as GVHD prophylaxis will be on day +1, day +3, and day +6
  Arms: Arm 2: Standard of Care

SUMMARY:
This randomized clinical trial will evaluate two approaches of GvHD prophylaxis; the standard of care GVHD prophylaxis regimen (methotrexate/calcineurin inhibitors) and post-transplant cyclophosphamide with calcineurin inhibitors for their efficacy as a new GVHD prophylaxis strategy.

DETAILED DESCRIPTION:
An open-label randomized clinical trial will be performed. Eligible patients are females and males, between 14 and 65 years undergoing allo-HCT for treatment of Acute Leukemia (AML or ALL). Patients must have a matching related peripheral blood stem cell donor. Patients from or referred to the KFSH&RC for allogeneic transplant consideration will be offered the opportunity to participate in this trial.

Treatment Description:

Patients will be randomized on one of the arms; an intervention or a standard of care arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Acute Leukemias (AML, ALL) in morphologic complete remission with or without hematologic recovery
* Patients must have a fully matched (8/8) related donor willing to donate peripheral blood stem cells and must meet institutional criteria for donation
* Planned Myeloablative conditioning regimen
* Cardiac function: ejection fraction at rest ≥ 50% by MUGA or TTE
* Estimated creatinine clearance greater than 50 mL/minute
* Pulmonary function: DLCO ≥ 50% (adjusted for hemoglobin), and FVC and FEV1 ≥ 50%
* Liver function: total bilirubin < 2x the upper limit of normal (unless elevated bilirubin is attributed to Gilbert's Syndrome) and ALT/AST < 2.5x the upper normal limit
* Signed informed consent

Exclusion Criteria:

* Karnofsky or Lansky Performance Score < 70%.
* Active disease
* Patients with uncontrolled bacterial, viral, or fungal infections
* Presence of fluid collection (ascites, pleural or pericardial effusion) that interferes with methotrexate clearance or makes methotrexate use contraindicated
* Patients seropositive for HIV-1 or -2
* Patients seropositive for HTLV-I or -II
* Patients with active Hepatitis B or C viral replication by PCR
* Women who are pregnant (positive serum or urine βHCG) or breastfeeding
* Females with childbearing potential (FCBP) or men who have sexual contact with FCBP unwilling to use effective forms of birth control or abstinence for one year after transplantation
* History of uncontrolled autoimmune disease or on active treatment
* Patients with prior malignancies, except resected non-melanoma skin cancer or treated cervical carcinoma in situ; cancer treated with curative intent ≥ 5 years previously will be allowed; cancer treated with curative intent < 5 years previously will not be allowed.

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
GRFS (GVHD-free/relapse-free survival) | One-year post-transplant
  Defined as the non-occurrence of a grade 3-4 acute GVHD, or systemic therapy-requiring chronic GVHD, or relapse, or death during the first post-transplant year.

SECONDARY OUTCOMES:
Acute Graft versus Host Disease (aGVHD) | 100 Day post transplant
  The probabilities of grade II-IV and III-IV acute GVHD will be determined. Acute GVHD will be graded according to Glucksberg and NIH 2014 criteria.
Chronic Graft versus Host Disease (cGVHD) | One year Post-transplant
  The cumulative incidence of systemic therapy-requiring chronic GVHD will be determined. Moderate and severe chronic GVHD will be defined per the NIH 2014 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Riad O El Fakih, MD, Principal Investigator — KFSH&RC; Mahmoud D Aljurf, MD, MPH, Principal Investigator — KFSH&RC; Marwan Y Shaheen, MD, Principal Investigator — KFSH&RC
Locations (1):
- King Faisal Specialist Hospital & Research Center, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No